CLINICAL TRIAL: NCT02240745
Title: New Three-dimensional Methods of Analysis for the Detection of Coronary Artery Disease by Dobutamine Stress Echocardiography
Acronym: 3-DSE
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 039/14; SNCTP 0761 (Other: KOFAM)
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease; Echocardiography, Stress
Keywords: Echocardiography, Stress; Echocardiography, Three-Dimensional; Coronary Artery Disease; Fractional Flow Reserve, Myocardial; Coronary Circulation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Patients with a suspicion of coronary heart disease
  Interventions: Other: Stress-echocardiography

INTERVENTIONS:
Other: Stress-echocardiography — Stress-echocardiography (incl dobutamin and atropin)

SUMMARY:
The investigators are going to recruit patients who have a scheduled elective coronary angiography and going to do a dobutamin stress echography (DSE) before the coronary examination. Next to a regular 2D-DSE, the investigators will perform an 3-dimensional DSE, incl ventriculography. In the interventional part (coronary angiography), they will measure each stenosis with fractional flow-reserve (FFR)and herewith graduate its stenosis severity.

DETAILED DESCRIPTION:
Background

Coronary heart disease is the leading cause of death worldwide. Non-invasive, radiation-free diagnostic needs further improvement. In this study, the investigators test the hypothesis that their method, which measures the myocardial deformation using 3D echocardiography is superior to previous ultrasound technologies with regard to diagnosis of stable coronary artery disease. The aim is establish an improved, non-invasive method to diagnose stable coronary artery disease.

Objective

The investigators want to investigate if a 3D-speckle-tracking is superior and more accurate in predicting hemodynamically significant coronary artery stenosis than predicted by 2D echocardiography? The reference variable for the hemodynamic significance of coronary artery stenosis is invasively measured by coronary flow reserve (CFR) in consideration of collateral flow (CFI).

Methods

This is a prospective observational study. The investigators will include 100 persons who are scheduled for an elective coronary angiography.

A regular 2D-stress echocardiography according to the international guidelines will be performed (incl. PLAX, SAX, 2CV, 4CV). The classification of regional wall motion abnormality is carried out according to the internationally recognized standards in 16 myocardial segments of the LV, with a grading of wall thickening (0 = dyskinetic, akinetic = 1, 2 = hypokinetic, 3 = normal). In addition, a 3D speckle tracking is performed after data transfer. To determine the functional relevance of any stenosis (reference method) a flow reserve in a maximum of two coronary arteries will be performed.

Test accuracy of 2D stress echocardiography and the new 3D method for detecting a significant stenosis (CFI <2) are then compared.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled elective coronary angiography
* Age >/= 18 years
* Written informed consent

Exclusion Criteria

* Age < 18 years
* Acute coronary syndrome
* Unstable angina pectoris
* Coronary 3-vessel disease
* Left-main artery affected
* Situation after myocardial infarction
* Coronary anomaly
* Situation after coronary bypass
* Congenital heart disease
* Pacemaker
* Any contraindication concerning stress-echo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 consecutive subjects referred to the Department of Cardiology for elective coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Area Strain in the affected coronary artery stenosis myocardial segments (Reference: Coronary flow reserve CFR) | After dobutamin-stress-echocardiography, PTCA will be performed within aprox.1-3hours
  Area Strain (%) by Echocardiography

SECONDARY OUTCOMES:
Area at Risk: Surface Area of site with reduced strain relative to the total LV-surface | After dobutamin-stress-echocardiography, PTCA will be performed within aprox.1-3hours
  Size of infarcted area according to the Area Strain (in % of total LV-surface)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano de Marchi, Senior consultant, Principal Investigator — Dept. of Cardiology, University Hospital of Bern, Bern
Locations (1):
- Dept of Cardiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Doucette JW, Corl PD, Payne HM, Flynn AE, Goto M, Nassi M, Segal J. Validation of a Doppler guide wire for intravascular measurement of coronary artery flow velocity. Circulation. 1992 May;85(5):1899-911. doi: 10.1161/01.cir.85.5.1899. PMID 1572046
- [Background] Traupe T, Gloekler S, de Marchi SF, Werner GS, Seiler C. Assessment of the human coronary collateral circulation. Circulation. 2010 Sep 21;122(12):1210-20. doi: 10.1161/CIRCULATIONAHA.109.930651. No abstract available. PMID 20855668
- [Background] Meuwissen M, Siebes M, Chamuleau SA, Tijssen JG, Spaan JA, Piek JJ. Intracoronary pressure and flow velocity for hemodynamic evaluation of coronary stenoses. Expert Rev Cardiovasc Ther. 2003 Sep;1(3):471-9. doi: 10.1586/14779072.1.3.471. PMID 15030274
- [Background] Varga A, Garcia MA, Picano E; International Stress Echo Complication Registry. Safety of stress echocardiography (from the International Stress Echo Complication Registry). Am J Cardiol. 2006 Aug 15;98(4):541-3. doi: 10.1016/j.amjcard.2006.02.064. Epub 2006 Jun 28. PMID 16893714